CLINICAL TRIAL: NCT03842488
Title: Multicenter, Open, Pilot Clinical Trial Aimed to Compare the Efficacy of RAL1200 QD vs DRV-cb 800-150 QD Both in Combination With TAF/FTC in Patients With HIV Infection and CD4 Count Under 200 Cells/microL
Brief Title: Raltegravir One Thousand Two Hundred vs Darunavir-cb in Immnunosupressed Patients: ROTDIP Study
Acronym: ROTDIP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIMHCSVIH-2017
Record Dates: First submitted 2018-12-19; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium; Tablets; Darunavir; Cobicistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RAL 1200 QD (Experimental): Start treatment with Raltegravir (RAL) 1200mg QD plus tenofovir alafenamide/emtricitabine (FTC/TAF)
  Interventions: Drug: Experimental: RAL QD
- DRV/cb (Active Comparator): Start treatment with Darunavir/Cobicistat (DRV/cb) 800-150mg QD plus tenofovir alafenamide/emtricitabine (FTC/TAF)
  Interventions: Drug: Active comparator: DRV/cb

INTERVENTIONS:
Drug: Experimental: RAL QD — Prescription of 2x RAL 600mg (1200MG) once daily
  Other Names: Raltegravir (RAL) 600mg Oral Tablet
  Arms: RAL 1200 QD
Drug: Active comparator: DRV/cb — Prescription of DARUNAVIR/COBICISTAT 800 Mg-150 Mg once daily
  Other Names: DARUNAVIR/COBICISTAT 800 Mg-150 Mg Oral Tablet
  Arms: DRV/cb

SUMMARY:
Multicenter, randomized, open label pilot clinical trial with two parallel arms aimed to compare the efficacy of Raltegravir (RAL) 1200mg QD vs Darunavir/Cobicistat (DRV-cb) 800-150mg QD both in combination with alafenamide/emtricitabine (TAF/FTC) in patients with Human Inmunodefficiency Virus (HIV) infection and CD4<200 cells/microL

DETAILED DESCRIPTION:
The trial consists of two parallel arms to study the therapeutic success of 48 weeks, tolerability, immunological recovery, persistence of treatment, safety and results reported by the subject in severely immunocompromised HIV infected patients (with an initial CD4 count <200 cells/μl) naive to antiretroviral therapy.

Included subjects will be randomized two to one (2:1) to RAL 1200mg QD plus FTC/TAF or DRV/cb (800-150mg) plus FTC/TAF.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18 years of age.
* HIV-1 infection.
* Naive to antiretroviral treatment.
* CD4 count at the beginning of the study <200 cells/μl.
* Estimated glomerular filtration ≥ 50 mL / min, according to the formula CKD-EPI.
* Grant Informed Consent in writing to participate in the study

Exclusion Criteria:

* Breastfeeding, pregnant or women in childbearing age who do not commit to maintain barrier contraceptive measures during the trial.
* Concomitant use of any drug with possible pharmacological interaction with the study drugs that it is advisable to "avoid" through the database for interactions at the University of Liverpool (www.hiv-druginteractions.org).
* Previous use of any antiretroviral for HIV infection.
* Resistance to the study drugs, or presence of any contraindication to use it. The inclusion in the study can be carried out before receiving the result of the resistance test. Once it is received, in case of presenting any mutation of resistance to drugs of the indicated regimen, the patient will be removed from the study and will be offered the best available treatment for their medical condition at that time.
* Therapies that include interferon, interleukin-2, cytotoxic chemotherapy or immunosuppressants at the entrance to the study.
* Current consumption of alcohol or other substances that at the discretion of the investigator may interfere with subject's treatment compliance.
* Subjects who currently participate in any other clinical trial using a research product, with the exception of studies in which the treatment studied has been stopped for more than 12 weeks.
* AIDS event in diagnosis of HIV infection or in the 3 months prior to the inclusion of the study.
* Suspected severe hepatopathy (grades B or C of the Child-Pugh classification), of any origin, according to the clinician.
* Any other clinical condition or previous treatment that, in the investigator's judgment, makes the subject unsuitable for the study or unable to comply with the dosage requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Compare efficacy of RAL 1200 mg QD versus DRV/cb 800-150 mg QD, both in combination with TAF/FTC | 48 weeks
  Number of patients that will improve when having raltegravir vs darunavir

SECONDARY OUTCOMES:
Virological failure | 48 weeks
  Number of patients in virological failure at week 48.
Compare the proportion of patients who interrupt the treatment for any reason | 48 weeks
  Number of patients that interrupt the treatment for any reason after 48 weeks.
Analyze change (percentage) in the number of CD4 lymphocytes | 48 weeks
  Percentage of change in the number of CD4 lymphocytes after 48 weeks.
Compare the proportion of patients with CD4>200 cells/μL at end of intervention | 48 weeks
  Compare the proportion of patients with CD4>200 cells/μL at end of intervention.
Percentage change in total cholesterol (TC) | 48 weeks
  Percentage of patients with change in total cholesterol (TC),
Percentage change in LDL and HDL cholesterol | 48 weeks
  Percentage of patients with change in LDL and HDL cholesterol
Percentage change in triglycerides | 48 weeks
  Percentage of patients with change the percentage change in triglycerides after 48 weeks
Percentage change in TC/HDL ratio | 48 weeks
  Percentage of patients with change in TC/HDL ratio
Change in Cardiovascular Risk 10-year predictive value (REGICOR). | 48 weeks
  Percentage of patients with change in Cardiovascular Risk 10-year predictive value (REGICOR).
Check GF modification using Chronic Kidney Disease Epidemiology (CKD-EPI) equation | 48 weeks
  Number of patiens with changes in glomerular filtration using Chronic Kidney Disease Epidemiology (CKD-EPI) equation.

IPD SHARING:
Plan to Share IPD: Undecided